CLINICAL TRIAL: NCT05025969
Title: Evaluation of the Incidence of NTRK Gene Fusion in Adult Brain Tumours
Acronym: NTRK Fusion
Status: Completed | Type: Observational
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Other Study IDs: COS-RGDS-2020-06-072
Record Dates: First submitted 2021-08-18; First posted 2021-08-30 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — The genomic analyses will be performed on tumour samples collected in routine practice during brain tumour removal surgery (glioma or brain metastasis) and the clinico-biological data will be collected from the medical records.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Glioma: (20 grade II gliomas, 20 grade III gliomas and 20 glioblastomas)
  Interventions: Other: Glioma data collection
- Brain metastasis: The "brain metastasis" cohort consists of 80 patients, including 30 patients for whom the matched primary tumour is available
  Interventions: Other: Brain metastasis data collection

INTERVENTIONS:
Other: Glioma data collection — Glioma data collection
  Groups: Glioma
Other: Brain metastasis data collection — Brain metastasis data collection
  Groups: Brain metastasis

SUMMARY:
This is a retrospective, mono centric, exploratory study to assess the incidence of a genomic alteration: NTRK gene fusion, in adult gliomas and brain metastases.

DETAILED DESCRIPTION:
Retrospective mono centric study of medical data (clinical, histological, molecular and imaging) from medical records and analysis of available excisional tissue samples.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female subject;
* Glioma or brain metastasis operated on in our institution, histologically confirmed (WHO classification 2016);
* Subject with a frozen tumour sample < 5 years old;
* Subject for whom all clinico-radiological data are available;
* Subject affiliated to a health insurance scheme;
* Subject who has been informed of the research and who has not indicated his opposition to the use of his medical data and who has signed a consent for the use of his tumour sample.

Exclusion Criteria:

* Patient under legal protection, guardianship or deprived of liberty by judicial or administrative decision
* Biological samples not available and/or in insufficient quantity for analysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients operated for glioma or brain metastasis.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2022-10-31 (Actual); Primary Completion 2023-02-08 (Actual); Study Completion 2023-02-08 (Actual)

PRIMARY OUTCOMES:
NTRK Fusion | through study completion, an average of 12 months
  Incidence of NTRK gene fusion identified by RNAseq in glioma and brain metastasis tumour samples.

SECONDARY OUTCOMES:
NTRK Fusion identification in brain metastasis and primary tumor | through study completion, an average of 12 months
  Incidence of NTRK gene fusion identified in matched pairs of brain metastasis and primary tumor;
Progression-free survival in patients with NTRK gene fusion | Month 6
  Progression-free survival in patients with NTRK gene fusion. Progression-free survival is defined as the time from the date of initial surgery to the date of diagnosis of progression. Progression will be defined according to the RANO criteria at 6 months
Progression-free survival in patients with NTRK gene fusion | Month 12
  Progression-free survival in patients with NTRK gene fusion. Progression-free survival is defined as the time from the date of initial surgery to the date of diagnosis of progression. Progression will be defined according to the RANO criteria at 12 months
Overall survival in patients with NTRK gene fusion. | through study completion, an average of 12 months
  Overall survival in patients with NTRK gene fusion. Overall survival is defined as the time from the date of initial surgery to the date of death (or the date of last news) of the patient.
Specific radiological criterion (T1) | through study completion, an average of 12 months
  Specific radiological criteria (T1) in patients with NTRK gene fusion in gliomas and brain metastases
Specific radiological criterion (T2) | through study completion, an average of 12 months
  Specific radiological criteria (T2) in patients with NTRK gene fusion in gliomas and brain metastases
Specific radiological criterion (FLAIR) | through study completion, an average of 12 months
  Specific radiological criteria (FLAIR) in patients with NTRK gene fusion in gliomas and brain metastases
Specific radiological criterion (perfusion) | through study completion, an average of 12 months
  Specific radiological criteria (perfusion) in patients with NTRK gene fusion in gliomas and brain metastases
Incidence of other genomic alterations | through study completion, an average of 12 months
  Incidence of other genomic alterations identified by RNAseq, associated with the incidence of NTRK gene fusion

CONTACTS AND LOCATIONS:
Overall Officials: Philippe METELLUS, MD PD, Principal Investigator — Hôpital Privé Clairval
Locations (1):
- Hôpital Privé Clairval, Marseille, France

IPD SHARING:
Plan to Share IPD: No